CLINICAL TRIAL: NCT00682500
Title: Calfactant Therapy for Direct Acute Respiratory Distress Syndrome & Direct Acute Lung Injury in Adults and Children
Brief Title: Calfactant for Direct Acute Respiratory Distress Syndrome
Acronym: CARDS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Expected mortality rates in placebo and treatment groups lower than predicted
Sponsor: Pneuma Pharmaceuticals Incorporated (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pneuma AR-06
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Pneumonia; Aspiration; Drowning; inhalation
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia; Drowning; Respiratory Aspiration | interventions — calfactant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Calfactant treatment
  Interventions: Drug: Calfactant
- 2 (Placebo Comparator)
  Interventions: Drug: Room Air (placebo)

INTERVENTIONS:
Drug: Calfactant — Intratracheal Instillation of 0.5 mL/cm of height of 60 mg/mL suspension in two aliquots at study entry. Repeat dosing 12 hours later if criteria are met.
  Other Names: PneumoSurf
  Arms: 1
Drug: Room Air (placebo) — Administration of 0.5 ml/cm height of air at study entry into the trachea. Repeat dosing at 12 hours if criteria are met
  Other Names: placebo
  Arms: 2

SUMMARY:
This study will determine if administration of an suspension of calfactant, a lung surfactant, intratracheally in patients with Direct Acute Respiratory Distress Syndrome within 48 hours of requiring mechanical ventilation can decrease the mortality in patients with lethal disease and shorten the course of respiratory failure in patients with sub-lethal disease.

DETAILED DESCRIPTION:
Recruitment limited to direct adult respiratory distress syndrome patients who have been intubated <48 hours. Origin of ARDS must be infectious pneumonia, aspiration of stomach contents, near drowning, smoke inhalation without pulmonary burn, inhaled industrial gas.

ELIGIBILITY:
Inclusion Criteria:

1. Respiratory failure due to diffuse infectious pneumonia, aspiration, near drowning, smoke inhalation or industrial gas
2. Less than 48 hours of mechanical ventilation
3. Informed consent

Exclusion Criteria:

1. Pre-existing lung disease
2. coma
3. limited therapeutic goals (do not resuscitate, etc.)
4. failure of another vital organ

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2008-05; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Mortality Rate | 90 days

SECONDARY OUTCOMES:
Duration of mechanical ventilation | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Willson, MD, Study Chair — Univeristy of Virginia Health Sciences Center; Jonathon Truwit, MD, Study Chair — University of Virginia Health Sciences Center
Locations (32):
- United States (18):
  - University of Florida, Gainesville, Florida
  - Florida Hospital and Florida Children's Hospital, Orlando, Florida
  - Northwestern University-Chicago, Chicago, Illinois
  - West Suburban Hospital Medical Center, Oak Park, Illinois
  - Peoria Pulmonary Associates/OSF St. Francis Hospital, Peoria, Illinois
  - Clarian Health, Inc/Methodist Hospital, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Creighton University, Omaha, Nebraska
  - Omaha Children's Hospital, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia Medical Center--Pediatrics, New York, New York
  - The Oregon Clinic, Portland, Oregon
  - Penn State University, Hershey, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - Uthscsa/Stvah, San Antonio, Texas
  - University of Virginia Health Science Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Canada (7):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Surrey Memorial Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - Kingston General Hospital, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
- Israel (2):
  - Haemek Medical Center, Jerusalem
  - Rabin Medical Center, Jerusalem
- New Zealand (2):
  - Auckland City Hospital, Auckland, Auckland
  - Starship Children's Hospital, Auckland, New Zealand
- South Korea (2):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Derived] Willson DF, Truwit JD, Conaway MR, Traul CS, Egan EE. The Adult Calfactant in Acute Respiratory Distress Syndrome Trial. Chest. 2015 Aug;148(2):356-364. doi: 10.1378/chest.14-1139. PMID 25855884